CLINICAL TRIAL: NCT05723497
Title: Supporting Local Agriculture Via Clinical Research: Human Studies With Elderberries to Improve Biomarkers of Obesity
Brief Title: Elderberries and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Patrick Solverson, Assistant Professor, Washington State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 18682
Record Dates: First submitted 2021-07-20; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Fuel Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderberry juice (Experimental): Participants will consume elderberry juice twice/day for 1-week.
  Interventions: Other: Elderberry juice
- Placebo beverage (Placebo Comparator): Participants will consume placebo beverage twice/day for 1-week.
  Interventions: Other: Placebo beverage

INTERVENTIONS:
Other: Elderberry juice — Participants will consume elderberry juice 1-week.
  Arms: Elderberry juice
Other: Placebo beverage — Participants will consume placebo for 1-week.
  Arms: Placebo beverage

SUMMARY:
Previous studies in humans indicate that anthocyanin-rich berries can positively alter fat oxidation and insulin sensitivity. This study will determine if this is also true with elderberries, which are a more concentrated source of anthocyanins compared to other commonly consumed berries.

ELIGIBILITY:
Inclusion Criteria:

Women and Men between 22 and 75 years of age with a body mass index of 25 kg/m2 or above.

Exclusion Criteria:

* Are not fully vaccinated against COVID-19 (at least 2-weeks out from final dose at time of staff meeting)
* Have a body mass index less than 25 kg/m2
* Are younger than 22 years of age, or older than 75 years of age
* Pregnant, lactating, or intending to become pregnant during the study period, or have given birth in the past year
* Known allergy or intolerance to elderberries
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease) or other metabolic disorders requiring a special diet that is not in accord with the diet behavior requested for this study
* Adherence to restrictive (vegetarian or vegan) or extreme (fad [ex. Ketogenic or Atkins] or quick weight loss/gain) diet patterns and unwillingness to consume a conventional, omnivorous diet and maintain body weight
* Habitual use of tobacco or marijuana (including vaping) products in the last 6 months
* Diagnosis or treatment of cancer in the past 3 years
* Crohn's disease or diverticulitis
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Use of certain medications (prescription or over-the-counter) that may interfere with the study objectives, including blood thinning medications
* Type 2 diabetes requiring the use of medication
* Fasting blood glucose > 125 mg/dL
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Substrate oxidation | 3.5 hours
  Participants will be monitored by a metabolic cart at rest and while walking
Glucose tolerance/insulin sensitivity | 3 hours
  Blood will be collected following a meal tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Physiology, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No